CLINICAL TRIAL: NCT04593108
Title: Study at Zagazig General Hospital
Brief Title: Misoprostol With or Without Letrozole in Treatment of Missed Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr.Dalia Mohammed Al Sayed Zaki (Other)
Collaborators: Benha University (Other)
Responsible Party: Sponsor-Investigator, Dr.Dalia Mohammed Al Sayed Zaki, Banha university, Benha University
Organization: Benha University (Other)
Other Study IDs: Treatment of missedmiscarriage
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Letrozole misoprostol: Group (A):
  A participant will receive three tablets of letrozole (Letrozole®, Technopharma) as a single dose, each tablet 2.5 mg (total dose 7.5 mg per day) on day One, then she took the second dose herself on day Two and will be told to bring back the empty pack. The third dose will be given on admission to hospital on day Three followed by 4 tablets of vaginal misoprostol (200 μg) (Cytotec®, Pfizer) soaked with saline every three hours for maximum two doses.then give antibiotics when abortion start
  Interventions: Device: Letrozole misoprostol
- Misoprostol,placebo: Group (B):
  A participant will receive three tablets of placebo as a single dose on day One, then she took the second dose herself on day Two and will be told to bring back the empty pack. The third dose will be given on admission to hospital on day Three followed by 4 tablets of vaginal misoprostol (200 μg) (Cytotec®, Pfizer) soaked with saline every three hours for maximum two doses.then give antibiotics when abortion start
  Interventions: Drug: Misoprostol, placebo

INTERVENTIONS:
Device: Letrozole misoprostol — Letrozole give pretreatment of abortion by misoprostol
  Groups: Letrozole misoprostol
Drug: Misoprostol, placebo — Give placebo pretreatment of abortion by misoprostol
  Groups: Misoprostol,placebo

SUMMARY:
Aim of study Compare the success rate of misoprostol with versus without letrozole as a pretreatment for medical termination of pregnancy during the first trimester.

Hypothesis:

Letrozole value as a pre-treatment medication for misoprostol in induction of abortion during the first trimester.

Research question:

Will letrozole- misoprostol protocol give better results than misoprostol- alone protocol in induction of abortion during the first trimester?

DETAILED DESCRIPTION:
Aim of the Work

Compare the success rate of misoprostol with versus without letrozole as a pretreatment for medical termination of pregnancy during the first trimester.

Hypothesis:

Letrozole value as a pre-treatment medication for misoprostol in induction of abortion during the first trimester.

Research question:

Will letrozole- misoprostol protocol give better results than misoprostol- alone protocol in induction of abortion during the first trimester?

Primary outcome:

Complete abortion (complete expulsion of products of conception with no need for curettage) within one week from the first dose of misoprostol.

Secondary outcome:

• Curettage (surgical evacuation of the products of conception)

* Incomplete abortion (retained products of conception).
* Considerable bleeding that necessitates immediate evacuation.

ELIGIBILITY:
Inclusion Criteria:

* Woman age more than 18 years old (age of legal consent).
* BMI ranges between 25 kg/m2 and 35 kg/m2.
* Gestational age of 63 days' gestation (or less).
* Missed abortion.
* Hemoglobin leve

Exclusion criteria:

* Woman age less than 18 years old.
* BMI less than 25 kg/m2 or more than 35 kg/m2.
* Gestational age more than 63 days' gestation.
* Molar pregnancy.
* Hemoglobin level less than 10 gm/dL.
* Fibroid uterus.
* Uterus with congenital anomalies.
* Previous attempts for induction of abortion in the current pregnancy.
* Coagulation defect i.e. coagulopathy.
* Contraindication for induction of abortion e.g. heart failure.
* Allergy to misoprostol or letrozole.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Study Settings:
  This clinical trial will be conducted in department of obstetrics and gynecology at Zagazig General Hospital during the period between January 2019 and June 2019.
  Study Population:
  The patients will be recruited from women attending outpatient clinic of obstetrics or the emergency room of Zagazig General Hospital.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
Complete abortion | 1week
  Complete abortion (complete expulsion of products of conception with no need for curettage) within one week from the first dose of misoprostol.

CONTACTS AND LOCATIONS:
Overall Officials: Zagazig General hospital, Ministry hospital, Principal Investigator — Zagazig general hospital
Locations (1):
- Dalia Mohammed Al Sayed Zaki, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee VCY, Ng EHY, Yeung WSB, Ho PC. Misoprostol with or without letrozole pretreatment for termination of pregnancy: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):317-323. doi: 10.1097/AOG.0b013e3182073fbf. PMID 21252745
- See also: Misoprostol with or without letrozole pretreatment for termination of pregnancy: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/21252745/
- Available data/document: Individual Participant Data Set — https://www.ncbi.nlm.nih.gov/m/pubmed/?term=Misoprostol+with+or+without+letrozole+in+treatment+of+missed+miscarriage+in+first+trimester+%5BJour%5D+AND+2018%5Bpdat%5D — Albrecht ED, Aberdeen GW, Pepe GJ, (2000). The role of estrogen in the maintenance of primate pregnancy. Am J Obstet Gynecol. 182:432-8. Albrecht ED, Robb VA, Pepe GJ, (2004). Regulation of placental vascular endothelial growth permeability factor expression and angiogenesis by estrogen during early baboon pregnancy. J Clin Endocrinol Metab. 89: